CLINICAL TRIAL: NCT06802666
Title: Short-course Radiotherapy(SCRT) Followed by Ivonescimab(AK112) and CAPOX as Neoadjuvant Therapy for Locally Advanced Rectal Cancer(LARC）: A Single-arm, Single-center, Exploratory, Phase II Clinical Study
Brief Title: Short-course Radiotherapy Followed by AK112 and CAPOX as Neoadjuvant Therapy for Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhenyu Lin, Director, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-IIT-C-S-0010
Record Dates: First submitted 2025-01-18; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Rectal Cancer; Neoadjuvant Therapy
MeSH Terms: interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: single arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCRT+AK112+chemotherapy (Experimental): short-course radiotherapy followed by sequential chemotherapy and AK112
  Interventions: Radiation: short-course radiotherapy; Drug: Ivonescimab; Drug: capecitabine; Drug: oxaliplatin; Procedure: TME surgery

INTERVENTIONS:
Radiation: short-course radiotherapy — Eligible subjects will receive short-course radiotherapy (SCRT). One week after the end of treatment, subjects continued to receive neoadjuvant chemotherapy combined with AK112 regimen for 6 cycles.
  Other Names: SCRT
Drug: Ivonescimab — AK112 20 mg/kg, intravenous infusion every 3 weeks (Q3W)
  Other Names: AK112
Drug: capecitabine — 1000mg/m2, bid, po, d1-14,q3w
Drug: oxaliplatin — 130mg/m2, ivgtt, d1,q3w
Procedure: TME surgery — The surgery was performed 1 week after the end of neoadjuvant therapy.

SUMMARY:
This study aims to evaluate the efficacy and safety of short-course radiotherapy followed by AK112 in combination with CAPOX as neoadjuvant therapy in patients with locally advanced rectal cancer

DETAILED DESCRIPTION:
Study includes a screening period (from the time the participant signs the informed consent form until the first treatment, not exceeding 21 days), treatment period (including full neoadjuvant therapy, surgery, and postoperative adjuvant treatment), and follow-up period (including safety follow-up and survival follow-up ).

Eligible subjects will receive short-course radiotherapy (SCRT). One week after the end of treatment, subjects continued to receive neoadjuvant chemotherapy combined with AK112 regimen for 6 cycles: AK112 20 mg/kg, intravenous infusion every 3 weeks (Q3W), plus CAPOX (capecitabine: 1000mg/m2, bid, po, d1-14, oxaliplatin: 130mg/m2, ivgtt, d1), Q3W.The surgery was performed 1 week after the end of neoadjuvant therapy.After surgery, the investigator conducts a pathological assessment of the surgical specimen for response evaluation. Then, there is a 30- and 90-day safety follow-up, and survival assessments are performed every 3 months to obtain survival information and collect new tumor treatment information until the death of the participant, withdrawal of informed consent, or the end of the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined this study, were able to complete the signing of the informed consent form, and had good compliance；
2. Age ≥18 years and ≤75 years, without gender restriction.
3. Histopathologically confirmed locally advanced rectal adenocarcinoma.
4. Participants who are not suitable for standard therapy due to intolerable toxicity, lack of standard therapy, or refusal of standard therapy.
5. Hematological parameters at baseline* (within 7 days prior to the first dose of study drug) must meet the following criteria: • Hemoglobin ≥90 g/L • Absolute neutrophil count (ANC) ≥1.5×10^9/L • Platelet count ≥100×10^9/L • Eosinophils ≤1.5×upper limit of normal (ULN). *Participants may not have received blood products (including red cell suspensions, plateletpheresis, cryoprecipitate), erythropoietin, or colony-stimulating factor supportive treatment within 7 days prior to blood sampling.
6. Serum biochemical tests at baseline (within 7 days prior to the first dose) must meet the following criteria: • Total bilirubin ≤1.5×ULN (if total bilirubin >1.5×ULN, direct bilirubin ≤ULN is acceptable for inclusion). • Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤3×ULN. • Serum creatinine ≤1.5×ULN or creatinine clearance (CCr) ≥45 mL/min, calculated using the Cockcroft-Gault formula (Appendix 4) using actual body weight. • Albumin ≥30 g/L.
7. Coagulation tests at baseline (within 7 days prior to the first dose) must meet the following criteria: • International normalized ratio (INR) ≤1.5×ULN (≤3×ULN if on stable anticoagulant therapy). • Partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤1.5×ULN (≤3×ULN if on stable anticoagulant therapy).
8. Urinalysis at baseline (within 7 days prior to the first dose) must meet the following criteria: urine protein (UPRO) <2+ or 24-hour urinary protein <1 g.
9. At least one measurable lesion according to RECIST v1.1 (solid tumors) criteria.
10. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
11. Expected survival ≥3 months.
12. Women of childbearing potential and male participants with female partners of childbearing potential must agree to use effective contraception throughout the treatment period and for 6 months after the end of treatment.

Exclusion Criteria:

1. Exclusion of patients not diagnosed with locally advanced rectal adenocarcinoma.
2. Participants who have previously received immunotherapy, including immune checkpoint inhibitors (such as anti-PD-1/L1 antibodies, anti-CTLA-4 antibodies, anti-TIGIT antibodies, anti-LAG-3 antibodies, etc.), immune checkpoint agonists (such as ICOS, CD40, CD137, GITR, OX40 antibodies, etc.), or any other treatments targeting tumor immunological mechanisms, such as immune cell therapy.
3. Pregnant or breastfeeding women, or women planning to become pregnant during the period from before the administration of the study drug, during treatment, or up to 6 months after the last dose.
4. Known history of active epilepsy, active central nervous system (CNS) metastases, spinal cord compression, carcinomatous meningitis, leptomeningeal disease, or new onset of brain or leptomeningeal metastases.
5. Significant cardiovascular diseases of clinical importance.
6. History of allergic constitution, asthma, or atopic dermatitis.
7. Participants with large pleural effusion or ascites.
8. Active autoimmune disease requiring systemic treatment (e.g., disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapies (e.g., thyroid hormone, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency) are not considered systemic treatment.
9. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
10. Participants known or suspected to be allergic to the investigational product or any of its excipients.
11. Participants with a history of significant toxicities associated with prior administration of immune checkpoint inhibitors or treatment with bevacizumab/pirfenidone-like agents that required permanent discontinuation of such treatment.
12. Participants with unresolved toxicity > Grade 1 related to any prior anticancer therapy (excluding persistent alopecia Grade 2, peripheral neuropathy, anemia, or hypomagnesemia).
13. Active uncontrolled bleeding or known bleeding diathesis, serious non-healing wounds, ulcers, or bone fractures, such as esophageal or gastric varices requiring immediate intervention (e.g., band ligation or sclerotherapy), or signs of portal hypertension where the Investigator believes the risk of bleeding is high.
14. Participants with a history of bowel obstruction (excluding those who have undergone curative surgery or have had complete resolution) or gastrointestinal perforation risk within 28 days prior to the first dose of this study (including but not limited to acute diverticulitis, abdominal abscess, peritoneal carcinomatosis, history of gastrointestinal perforation and/or fistula within 6 months prior to study entry).
15. Current or recent (within 6 months) major gastrointestinal diseases or conditions in participants, including:

    1. Clinically significant history of gastrointestinal bleeding.
    2. Active peptic ulcer disease.
    3. ≥Grade 2 diarrhea occurring within 2 weeks prior to the first dose of the study drug.
16. Participants who have received chemotherapy, small molecule inhibitors, immunotherapy (such as interleukins, interferons, or thymosin) for cancer treatment within 28 days before this study, or traditional Chinese medicine with anti-cancer indications within 14 days prior to dosing.
17. Known positive HIV test result, active hepatitis B, hepatitis C (HCV), tuberculosis, or a history of infection with these diseases.
18. Serious/active/uncontrolled infection or infection requiring systemic intravenous antibiotics, or fever of unknown origin (>38°C) within 2 weeks prior to the first dose of the study drug.
19. Diagnosis of another malignancy within 5 years prior to the first dose, except for cases such as adequately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or carcinoma in situ that has been surgically resected, as well as localized prostate cancer or papillary thyroid cancer post-radical surgery.
20. Participants who have received radical radiotherapy within 3 months prior to this study; palliative radiotherapy is allowed if administered at least 2 weeks prior to dosing and the radiation dose is consistent with local standards for palliative care.
21. Presence of any medical condition, therapy, laboratory abnormality, or history of drug abuse, or current evidence thereof, which in the opinion of the investigator might jeopardize the safety of the participant, interfere with obtaining informed consent, affect the participant's compliance, or impact the assessment of the safety of the study drug.
22. Patients whom the investigator deems unsuitable for participation in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate (pCR) | though 19 weeks neoadjuvant treatment，after surgery completed
  Pathological complete response will be made based on assessment of the surgical specimen at the primary treatment site，the absence of any viable tumor cells in the resected primary tumor specimen and all regional lymph node samples.

SECONDARY OUTCOMES:
3-years Event-Free Survival rate | 3 years
  from the start of randomized treatment assignment until the occurrence of a predefined event
OS | From date of randomization until date of death from any cause，up to 3 years
  To compute the length between end of treatment and death
R0 resection rate | From date of surgry，up to 1month
  The rate of negative margin microscopically
AE | up to 3 years
  To assess the result from inspection paper during the trail，adverse events (AEs) were graded according to the NCl CTCAE version 5.0
30-day postoperative mortality rates | 30 days post surgery
  30-day mortality rate after rectal cancer surgery
Surgical complications | After surgery，up to 3years
  Possible complications that may occur after rectal cancer surgery
90-day postoperative mortality rates | 90 days post surgery
  90-day mortality rate after rectal cancer surgery
length of hospital stay | through study completion, an average of 1 year
  Length of Postoperative Hospital Stay

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, MD, Study Director — Union Hospital affiliated to Tongji Medical College of Huazhong University ofScience and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Hubei, China

IPD SHARING:
Plan to Share IPD: No